CLINICAL TRIAL: NCT06543836
Title: ctDNA-guided Treatment of an Anti-angiogenic TKI Combined With a PD-1 Inhibitor for Advanced pMMR/MSS Colorectal Cancer Failed With Standard Therapy: a Randomized Controlled Phase 2 Clinical Trial
Brief Title: ctDNA-guided Treatment of TKI Plus PD-1 Inhibitor for Advanced pMMR/MSS Colorectal Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, AIPING ZHOU, Professor, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCC4663
Record Dates: First submitted 2024-07-15; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — sintilimab; Immune Checkpoint Inhibitors; HMPL-013; regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PD-1 inhibitor+Tyrosine kinase inhibitor(TKI) (Experimental): PD-1 inhibitor: Sintilimab 200mg, d1, TKI: Fruquintinib 5mg Qd, d1-14, Q3w. Efficacy assessment every 2 cycles.
  Interventions: Drug: Sintilimab; Drug: Fruquintinib
- Tyrosine kinase inhibitor(TKI) (Active Comparator): The treatment regimen consists of the following options:
  Option 1: Fruquintinib 5mg Qd, d1-21, Q4w, and efficacy assessment every 1.5 months.
  Option 2: Regorafenib 160mg Qd, d1-21, Q4w, and efficacy assessment every 1.5 months.
  Interventions: Drug: Fruquintinib or Regorafenib

INTERVENTIONS:
Drug: Sintilimab — Sintilimab 200mg, d1, with a treatment cycle of 21 days, and efficacy assessment every 2 cycles.
  Other Names: PD-1 inhibitor
  Arms: PD-1 inhibitor+Tyrosine kinase inhibitor(TKI)
Drug: Fruquintinib or Regorafenib — The treatment regimen consists of the following options:
  Option 1: Fruquintinib 5mg Qd, d1-21, Q4w, and efficacy assessment every 1.5 months.
  Option 2: Regorafenib 160mg Qd, d1-21, Q4w, and efficacy assessment every 1.5 months.
  Other Names: TKI
  Arms: Tyrosine kinase inhibitor(TKI)
Drug: Fruquintinib — Fruquintinib 5mg Qd, d1-14, with a treatment cycle of 21 days, and efficacy assessment every 2 cycles.
  Other Names: TKI
  Arms: PD-1 inhibitor+Tyrosine kinase inhibitor(TKI)

SUMMARY:
The efficacy of combining TKI with PD-1 inhibitor in the treatment of advanced MSS/pMMR colorectal cancer with low levels of maxVAF in peripheral blood ctDNA failed with standard treatment was assessed, compared to standard treatment as chosen by researchers.

DETAILED DESCRIPTION:
This study is a prospective, randomized phase II controlled trial. It will include patients with histologically confirmed advanced metastatic pMMR/MSS colorectal adenocarcinoma, who have failed with treatment with fluoropyrimidine (5-fluorouracil or capecitabine), oxaliplatin, irinotecan plus bevacizumab/cetuximab (left-side RAS/BRAF wild-type) and whose peripheral blood ctDNA test shows a maxVAF level lower than 6.5%. Patients will be randomly assigned to receive a TKI + a PD-1 inhibitor (primarily fruquintinib combined with sintilimab) or standard later-line treatment options (regorafenib or fruquintinib monotherapy, at the discretion of the investigator) until disease progression, death, intolerable adverse events, or withdrawal of informed consent.

ELIGIBILITY:
Inclusion Criteria:

1. Age range between 18 and 80 years old.
2. ECOG performance status of 0 or 1.
3. Histologically confirmed advanced or recurrent colorectal adenocarcinoma.
4. Confirmed normal expression of mismatch repair proteins (pMMR) by immunohistochemistry or microsatellite stable (MSS) by PCR/next-generation sequencing.
5. Blood ctDNA maxVAF <6.5% as detected by NGS. blood samples of 8-10ml are to be collected from a qualified testing company for analysis.
6. Metastatic colorectal cancer that has failed with previous treatment with fluoropyrimidine (5-fluorouracil or capecitabine), oxaliplatin, irinotecan plus bevacizumab/cetuximab (left-side RAS/BRAF wildtype).
7. At least 28 days since the last systemic therapy (oral fluoropyrimidine ≥ 14 days), with the option of receiving palliative radiation therapy to limited areas if completed more than 3 weeks prior.
8. At least one measurable lesion according to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST V1.1).
9. Expected survival of at least 3 months.
10. Adequate organ and bone marrow function, with laboratory values within the following limits within 7 days before enrollment:

    1. Complete blood count: Absolute neutrophil count (ANC) ≥1.5×10^9/L, Platelet count (PLT) ≥100×10^9/L, Hemoglobin (HGB) ≥9.0 g/dL.
    2. Liver function: Total bilirubin (TBIL) ≤1.5× upper limit of normal (ULN), Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5× ULN, or ≤5× ULN in the presence of liver metastasis.
    3. Kidney function: Serum creatinine (Cr) ≤1.5×ULN, or creatinine clearance ≥50ml/min, Urinalysis showing urine protein <2+, for patients with baseline urine protein ≥2+, 24-hour urine protein collection should show <1g.
    4. Coagulation function: International normalized ratio (INR) and activated partial thromboplastin time (APTT) ≤1.5 times ULN.
11. Normal electrocardiogram, left ventricular ejection fraction (LVEF) ≥50%.
12. No history of other malignancies, except for cured cervical carcinoma in situ, non-melanoma skin cancer, non-invasive bladder tumors, non-invasive lung cancer, or malignant tumors with continuous disease-free survival of ≥5 years following surgical resection.
13. Negative pregnancy test for women of childbearing potential, and willingness to use effective contraception during the clinical trial period.
14. Voluntary participation in the clinical trial with informed consent provided.

Exclusion Criteria:

1. Patients with a history of prior treatment with fruquintinib or similar small molecule oral targeted drugs primarily aimed at anti-angiogenesis (including marketed or investigational drugs).
2. Patients with a history of prior treatment with other PD-1/PD-L1/CTLA-4 antibody therapies or other immunotherapies targeting PD-1/PD-L1/CTLA-4.
3. Patients who experienced severe hypersensitivity reactions after monoclonal antibody administration in the past.
4. Patients with any active autoimmune disease or a history of autoimmune diseases (such as, but not limited to: autoimmune hepatitis, interstitial pneumonia, enteritis, vasculitis, nephritis, and patients requiring bronchodilators for medical intervention for asthma cannot be included). however, the following patients are allowed to be included: patients with vitiligo, psoriasis, alopecia that do not require systemic treatment, well-controlled type I diabetes, and hypothyroidism with normal thyroid function under replacement therapy.
5. Patients who require immunosuppressive agents, systemic corticosteroids, or absorbable local steroid therapy for achieving immunosuppression (dose >10mg/day prednisone or equivalent) and are still on continued therapy within 2 weeks of initial dosing.
6. Patients with various factors affecting oral drug intake (such as dysphagia, post-gastrointestinal surgery, chronic diarrhea, and intestinal obstruction).
7. Patients with uncontrollable pleural effusion, pericardial effusion, or ascites requiring repeated drainage.
8. Patients with any signs or history of bleeding diathesis regardless of severity, patients who experienced any bleeding event ≥CTCAE Grade 3 within 4 weeks before initial dosing, or patients with unhealed wounds, fractures, active peptic ulcers, ulcerative colitis, or other gastrointestinal diseases with active bleeding or other conditions deemed by the investigator to potentially cause severe gastrointestinal bleeding or perforation.
9. Patients with known brain metastases with a history of organ transplantation.
10. Patients who received approved or investigational anti-tumor treatments within 4 weeks before the start of the study, including but not limited to chemotherapy, surgery, radiotherapy (within 3 weeks), biologically targeted therapy, interventional therapy, immunotherapy, and traditional Chinese medicine treatment for cancer (as per the indications in the traditional Chinese medicine instructions, participants can be included after a 2-week washout period) (Note: oral fluoropyrimidine drugs for less than 14 days, patients with adverse events from previous treatments, excluding alopecia, not recovered to ≤CTCAE Grade 1).
11. Patients vaccinated with preventive or attenuated vaccines within 4 weeks before the first dose.
12. Patients with any severe and/or uncontrolled diseases, including:

    1. patients with suboptimal blood pressure control (systolic blood pressure ≥150 mmHg, diastolic blood pressure ≥90 mmHg).
    2. patients who had thrombotic events, cerebrovascular accidents, myocardial infarctions, ≥Grade 2 congestive heart failure, or requiring treatment for arrhythmias (including QTc ≥480ms) within 6 months before the first dose.
    3. patients with active or uncontrolled severe infections (≥CTCAE Grade 2 infections), tuberculosis patients.
    4. patients with a clinically significant history of liver disease, including viral hepatitis, known carriers of hepatitis B virus (HBV) must exclude active HBV infection, i.e., HBV DNA positive (>1 × 10^4 copies/mL or >2000 IU/mL), known hepatitis C virus infection (HCV) and HCV RNA positive (>1 × 10^3 copies/mL), or other decompensated liver diseases, chronic hepatitis requiring antiviral treatment.
    5. HIV positive.
    6. poorly controlled diabetes (fasting blood sugar ≥CTCAE Grade 2).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
PFS | Up to 2 years
  Progression-free survival

SECONDARY OUTCOMES:
OS | Up to 2 years
  Overall survival
ORR | Up to 2 years
  Objective response rate
DCR | Up to 2 years
  Disease control rate

CONTACTS AND LOCATIONS:
Overall Officials: Aiping Zhou, M.D., Principal Investigator — Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College
Locations (1):
- National Cancer Center/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No